CLINICAL TRIAL: NCT03144830
Title: Exoskeleton Use in Acute Rehab Post Spinal Cord Injury; a Safety and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Chester Ho, MD, Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EKSO22214
Record Dates: First submitted 2016-04-20; First posted 2017-05-09 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exoskeleton Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overground walking program (Experimental): Study participant will be involved in an indoor, overground walking program using an exoskeleton wearable walking device under the supervision of a physiotherapist.
  Interventions: Device: Exoskeleton

INTERVENTIONS:
Device: Exoskeleton — This is an open study and so all participants involved with be using the exoskeleton to determine the safety and feasibility of its use during the acute rehabilitation phase.
  Other Names: Ekso GT

SUMMARY:
This study will examine the safety and feasibility of using an exoskeleton in subjects who are less than 6 months post spinal cord injury (SCI).

DETAILED DESCRIPTION:
Study participants with acute SCI (<6 months post injury) will be involved in an indoor, overground walking program.

Locomotor training will include 90 minute sessions (including time to don and doff the device) for 30 training hours (90 minutes, 2-3 times weekly for 8 weeks.)

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 15 and older with acute SCI (<6 months post) Etiology of SCI can be traumatic or non traumatic Includes motor complete (AIS A,B) and motor incomplete (AIS C,D) at C7 or below.

Participants must be able to follow 2 step commands Participants must be deemed medically stable by responsible physician or physiatrist

* Spine considered stable by surgeon
* Surgical wound is approximated and surrounding tissue appears healthy
* Participant does not require supplemental Oxygen
* Participant is able to have any IV or other lines disconnected.

Must meet manufacturer's requirements for use of Ekso GT:

Exclusion Criteria:

* Range of motion (ROM) restrictions that would prevent a patient from achieving a normal, reciprocal gait pattern, or would restrict a patient from completing normal sit-to-stand or stand-to-sit transitions Spinal instability Untreated deep vein thrombosis (DVT) Decreased standing tolerance due to orthostatic hypotension Significant osteoporosis that prevents safe standing or may increase the risk of fracture caused by standing or walking Uncontrolled spasticity - score of 3 or higher on modified Ashworth Scale Uncontrolled Autonomic Dysreflexia (AD) Skin integrity issues on contact surfaces of the device or on surfaces that would prohibit sitting (sacrum, greater trochanter, proximal tibia)

Upper leg length discrepancy greater than half an inch (> .5") or lower leg discrepancy greater than three-quarters of an inch (>.75") Cognitive impairments resulting in motor planning or impulsivity concerns Pregnancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline cardiorespiratory status throughout each of the 25 sessions | Every 15 minutes during each training session including: pre and post initial stand, at 15 minute intervals during training and at the end of each of the 25 total sessions, on average of 2 months
  Blood pressure, heart rate and peripheral oxygen saturation and will be used to identify any cardiovascular issues of orthostatic hypotension or autonomic dysreflexia.

SECONDARY OUTCOMES:
Skin integrity | At the beginning and end of each training session for 25 sessions, on average of 2 months
  A visual inspection of areas of significant weight bearing and skin/machine interface will take place at the beginning and end of each training session to monitor for skin breakdown or compromise.
Falls | From onset to cessation of each training session for 25 sessions, on average of 2 months
  Any incidence of falls will be recorded and the participant will be evaluated for injury by unit medical staff or on site emergency staff if warranted.
Pain visual analogue scale | At the beginning and end of each training session for 25 sessions, on average of 2 months
  Participants draw an intersecting line on a 10 cm line (scale) in order to rate their amount of subjective pain. The distance on the 10 cm line is measured from the left side (no pain) and turned into a numerical value.
Borg scale of perceived exertion | At the beginning, mid point (30 min) and end (60 min) of each training session for 25 sessions, on average of 2 months
  Subjects are shown the Borg scale of perceived exertion and are asked to choose the number/descriptor that best aligns with their current level of exertion at 0, 30 and 60 minutes.
10 meter walk test | Training sessions 1, 13 and 25 out of the 25 total sessions, on average of 2 months
  Time in seconds it takes a subject to walk a distance of 10 meters.
6 minute walk test | Training sessions 1, 13 and 25 of the 25 total sessions, on average of 2 months
  Total distance a participant is able to walk in 6 minutes will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Chester Ho, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No